CLINICAL TRIAL: NCT07029438
Title: Clinical Study to Evaluate the Comparative Efficacy of Floss, Essential Oil Mouthwashes, and an Alcohol-free CPC+Zn Mouthwash in Reducing Dental Plaque and Gingivitis
Brief Title: Comparative Efficacy of Floss and Essential Oil/CPC+Zn Mouthwashes in Reducing Dental Plaque and Gingivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRO-2025-FlossRinse-PG-GJ
Record Dates: First submitted 2025-05-29; First posted 2025-06-19 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-06

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Mouthwashes; Dental Devices, Home Care; Toothpastes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Brushing (Placebo Comparator): Subjects will brush their teeth in their usual manner for 1 timed minute twice daily with the toothbrush and toothpaste provided. They will apply the toothpaste on the full length of the toothbrush. This arm will be the negative control arm (placebo comparator).
  Interventions: Device: Toothbrush; Drug: Toothpaste
- Brushing and Flossing (Experimental): Subjects will brush their teeth in their usual manner for 1 timed minute twice daily with the toothbrush and toothpaste provided. They will apply the toothpaste on the full length of the toothbrush. Subjects will floss their teeth after their first brushing instance of the day per instructed method from the study site.
  Interventions: Device: Floss; Device: Toothbrush; Drug: Toothpaste
- Brushing and Rinsing A (Experimental): Subjects will brush their teeth in their usual manner for 1 timed minute twice daily with the toothbrush and toothpaste provided. They will apply the toothpaste on the full length of the toothbrush. After both brushing instances, subjects will rinse full strength with 20 mL of Mouthwash A for 30 timed seconds.
  Interventions: Drug: Mouthwash; Device: Toothbrush; Drug: Toothpaste
- Brushing and Rinsing B (Experimental): Subjects will brush their teeth in their usual manner for 1 timed minute twice daily with the toothbrush and toothpaste provided. They will apply the toothpaste on the full length of the toothbrush. After both brushing instances, subjects will rinse full strength with 20 mL of Mouthwash B for 30 timed seconds.
  Interventions: Drug: Mouthwash; Device: Toothbrush; Drug: Toothpaste
- Brushing and Rinsing C (Experimental): Subjects will brush their teeth in their usual manner for 1 timed minute twice daily with the toothbrush and toothpaste provided. They will apply the toothpaste on the full length of the toothbrush. After both brushing instances, subjects will rinse full strength with 20 mL of Mouthwash C for 30 timed seconds.
  Interventions: Drug: Mouthwash; Device: Toothbrush; Drug: Toothpaste

INTERVENTIONS:
Drug: Mouthwash — Antiplaque/Antigingivitis Mouthwash
  Arms: Brushing and Rinsing A; Brushing and Rinsing B; Brushing and Rinsing C
Device: Floss — Dental Floss
  Arms: Brushing and Flossing
Device: Toothbrush — Soft bristled, manual toothbrush
Drug: Toothpaste — Sodium Monofluorophosphate 0.76 % (0.15% w/v fluoride ion) toothpaste

SUMMARY:
The objective of this clinical research study is to evaluate the efficacy of floss to an essential oil alcohol-containing mouthwash, an essential oil alcohol-free mouthwash, and a CPC+Zn alcohol-free mouthwash in reducing dental plaque and gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers at least 18 years of age and in general good health.
* Willing and able to understand and sign the informed consent form.
* Whole mouth mean MGI ≥1.95, whole mouth mean TPI≥1.95, and ≥10% bleeding sites
* Be willing to conform to the study protocol and procedures.
* No sites with probing depth >4 mm.
* Minimum of 20 natural teeth with scorable facial and lingual surfaces

Exclusion Criteria:

* Medical condition which requires premedication prior to dental visits/procedure.
* Known history of allergy to personal care/consumer products or their ingredients, relevant to any ingredients in the test products as determined by the study examiner.
* Active disease of the hard oral tissues.
* Significant oral soft tissue pathology, excluding plaque-induced gingivitis.
* Moderate to severe periodontitis (stages II-IV) per the EFP S3 guidelines.
* Subjects with fixed or removable orthodontic appliances or removable partial dentures.
* Dental prophylaxis within 30 days prior to study start.
* Use of antibiotics, antimicrobial drugs, anti-inflammatory drugs, or anticoagulant therapies within 30 days prior to study start.
* Use of chemotherapeutic oral care products within two weeks prior to study start.
* Participation in any other clinical study within 30 days prior to enrollment into this study.
* Subjects who must receive dental treatment during the study dates.
* Immunocompromised individuals (HIV, AIDS, immunosuppressive drug therapy).
* Use of smokeless tobacco, vaping, or e-cigarettes or suspected substance abuse.
* Current smokers (if former smoker, should have stopped at least 1 month prior to Visit 1)
* Pregnant or lactating subjects, or subjects planning to become pregnant during the course of the study.
* Medical condition which prohibits not eating/drinking or chewing gum for four (4) hours prior to your scheduled visits;
* Subjects who have an infectious disease and/or other blood borne diseases (Hepatitis series, HIV, tuberculosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Interproximal mean Modified Gingival Index (MGI) | 12 weeks
  MGI will be visually assessed for six sites for each graded tooth (mesiofacial, facial, distofacial, mesiolingual, lingual, distolingual). Interproximal MGI includes the mesiofacial, distofacial, mesiolingual, and distolingual sites. Higher scores indicate a worse outcome, per below.
  0 = no inflammation; no redness
  1. = mild inflammation; slight changes in color and texture, but not in all portions of gingival marginal or papillary
  2. = mild inflammation; slight changes in color and texture in all portions of gingival margin or papillary
  3. = moderate inflammation; bright surface inflammation, erythema, edema, and/or hypertrophy of gingival marginal or papillary
  4. = severe inflammation; erythema, edema, and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion, or ulceration

SECONDARY OUTCOMES:
Whole Mouth mean Modified Gingival Index (MGI) | 1, 4, and 12 weeks
  MGI will be visually assessed for six sites for each graded tooth (mesiofacial, facial, distofacial, mesiolingual, lingual, distolingual). Whole Mouth MGI includes all six sites. Higher scores indicate a worse outcome, per below.
  0 = no inflammation; no redness
  1. = mild inflammation; slight changes in color and texture, but not in all portions of gingival marginal or papillary
  2. = mild inflammation; slight changes in color and texture in all portions of gingival margin or papillary
  3. = moderate inflammation; bright surface inflammation, erythema, edema, and/or hypertrophy of gingival marginal or papillary
  4. = severe inflammation; erythema, edema, and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion, or ulceration
Interproximal mean Turesky Modification of the Quigley-Hein Plaque Index (TPI) | 1, 4, and 12 weeks
  Dental plaque will be assessed at six sites for each graded tooth (mesiofacial, facial, distofacial, mesiolingual, lingual, distolingual) and scored as follows:
  0=No plaque
  1. Separate flecks of plaque at the cervical margin
  2. A thin, continuous band of plaque (up to 1 mm) at the cervical margin
  3. A band of plaque wider than 1 mm, but covering less than 1/3 of the side of the crown of the tooth
  4. Plaque covering at least 1/3, but less than 2/3 of the side of the crown of the tooth
  5. Plaque covering 2/3 or more of the side of the crown of the tooth
  Interproximal mean includes mesiofacial, distofacial, mesiolingual, and distolingual sites. Higher scores indicate a worse outcome, per above.
Whole Mouth mean Turesky Modification of the Quigley-Hein Plaque Index (TPI) | 1, 4, and 12 weeks
  Dental plaque will be assessed at six sites for each graded tooth (mesiofacial, facial, distofacial, mesiolingual, lingual, distolingual) and scored as follows:
  0=No plaque
  1. Separate flecks of plaque at the cervical margin
  2. A thin, continuous band of plaque (up to 1 mm) at the cervical margin
  3. A band of plaque wider than 1 mm, but covering less than 1/3 of the side of the crown of the tooth
  4. Plaque covering at least 1/3, but less than 2/3 of the side of the crown of the tooth
  5. Plaque covering 2/3 or more of the side of the crown of the tooth
  Whole Mouth mean includes all six sites. Higher scores indicate a worse outcome, per above.
Interproximal mean Expanded Bleeding Index (EBI) | 1, 4, and 12 weeks
  EBI will be assessed at six sites for each graded tooth (mesiofacial, facial, distofacial, mesiolingual, lingual, distolingual) by engaging a probe 1 mm into the gingival crevice and applying moderate pressure whilst sweeping from interproximal to interproximal along the sulcular epithelium. Interproximal mean includes mesiofacial, distofacial, mesiolingual, and distolingual sites. A higher score indicates a worse outcome, per below.
  0 = no bleeding after 30 seconds
  1. = bleeding upon probing after 30 seconds
  2. = immediate bleeding observed
Whole Mouth Expanded Bleeding Index (EBI) | 1, 4, and 12 weeks
  EBI will be assessed at six sites for each graded tooth (mesiofacial, facial, distofacial, mesiolingual, lingual, distolingual) by engaging a probe 1 mm into the gingival crevice and applying moderate pressure whilst sweeping from interproximal to interproximal along the sulcular epithelium. Whole Mouth mean includes all six sites. A higher score indicates a worse outcome, per below.
  0 = no bleeding after 30 seconds
  1. = bleeding upon probing after 30 seconds
  2. = immediate bleeding observed
Interproximal mean Bleeding on Probing (BOP) | 12 weeks
  Bleeding on probing will be assessed at six sites for each graded tooth (mesiofacial, facial, distofacial, mesiolingual, lingual, distolingual) and scored as 1 = yes bleeding, 0 = no bleeding. Interproximal mean includes mesiofacial, distofacial, mesiolingual, and distolingual sites. A higher score indicates a worse outcome.
Whole Mouth mean Bleeding on Probing (BOP) | 12 weeks
  Bleeding on probing will be assessed at six sites for each graded tooth (mesiofacial, facial, distofacial, mesiolingual, lingual, distolingual) and scored as 1 = yes bleeding, 0 = no bleeding. Whole Mouth mean includes all six sites. A higher score indicates a worse outcome.
Interproximal mean Probing Depth (PD) | 12 weeks
  Probing depth will be measured at six sites for each graded tooth (mesiofacial, facial, distofacial, mesiolingual, lingual, distolingual) using a calibrated periodontal probe to ensure precision and consistency. Interproximal mean includes mesiofacial, distofacial, mesiolingual, and distolingual sites.
  Measurements will be recorded to the nearest millimeter, with particular attention to maintaining gentle and consistent pressure to avoid measurement variability. Larger measurements indicate a worse condition.
Whole Mouth mean Probing Depth (PD) | 12 weeks
  Probing depth will be measured at six sites for each graded tooth (mesiofacial, facial, distofacial, mesiolingual, lingual, distolingual) using a calibrated periodontal probe to ensure precision and consistency. Interproximal mean includes mesiofacial, distofacial, mesiolingual, and distolingual sites.
  Measurements will be recorded to the nearest millimeter, with particular attention to maintaining gentle and consistent pressure to avoid measurement variability. Larger measurements indicate a worse condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, MPA, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF, CSR